CLINICAL TRIAL: NCT01792609
Title: Minimize Implants Maximize Outcomes (MIMO) Clinical Trial
Brief Title: Min Implants Max Outcomes Clinical Trial
Acronym: MIMOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other); Texas Scottish Rite Hospital for Children (Other); Johns Hopkins University (Other); University of Rochester (Other); Washington University School of Medicine (Other); Children's Hospital Colorado (Other); Mayo Clinic (Other); University of Iowa (Other); Norton Leatherman Spine Center (Other); Children's Hospital of Philadelphia (Other); St. Justine's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1208M18202
Record Dates: First submitted 2013-01-22; First posted 2013-02-15 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Scoliosis; Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Cobb Angle; Screw Density; Outcomes Measures
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maximum Number of Screws (Active Comparator): Once enrolled and consented, patients with Lenke 1A curves will be randomized to a high- or low-density screw cohort. The high-density pattern will be designated as ≥ 1.8 implants per level fused. The low density pattern will be ≤ 1.4 screws per level fused. At least 75% of the implants must be pedicle screws for both cohorts.
  Interventions: Procedure: Maximum Number of Screws
- Minimum Number of Screws (Active Comparator): Once enrolled and consented, patients with Lenke 1A curves will be randomized to a high- or low-density screw cohort. The high-density pattern will be designated as ≥ 1.8 implants per level fused. The low density pattern will be ≤ 1.4 screws per level fused. At least 75% of the implants must be pedicle screws for both cohorts.
  Interventions: Procedure: Minimum Number of Screws

INTERVENTIONS:
Procedure: Maximum Number of Screws — The tools used for this arm of study are FDA approved with section 510 (k) K122433. These screws are regularly used in all procedures pertaining to Cobb angle correction surgeries outside of the context of this study.
  Other Names: Pedicle Screw Spinal System
  Arms: Maximum Number of Screws
Procedure: Minimum Number of Screws — The tools used for this arm of study are FDA approved with section 510 (k) K122433. These screws are regularly used in all procedures pertaining to Cobb angle correction surgeries outside of the context of this study.
  Other Names: Pedicle Screw Spinal System
  Arms: Minimum Number of Screws

SUMMARY:
Objectives Primary objective: Determine if there is a clinically significant difference in percent Cobb curve correction in a low- vs. high-implant density cohort through a prospective randomized controlled trial.

Design and Outcomes Randomized clinical trial of equivalence to test the efficacy and safety of low vs. high implant density instrumentation for spine deformity surgery in AIS patients with Lenke IA curve patterns.

Interventions and Duration Intervention: low-implant density group or high-implant density group. Duration: 2 years. Sample Size and Population Target population: 10 to 17 years old with AIS who will undergo instrumented spinal fusion. Sample size needed (power = 90%) is 174 subjects with 87 in each group.

DETAILED DESCRIPTION:
The MIMO Study Group proposes to conduct a prospective randomized controlled trial in order to determine whether a low implant density cohort has equivalent clinical and radiographic results to a high implant density cohort. This study is proposed as a trial of equivalence. The null hypothesis is that significant differences exist in percent major Cobb angle correction between high- and low-implant density cohorts for Lenke 1A curve types, the most common scoliotic curve pattern (73). Consecutive qualifying patients will be screened and enrolled by high-volume spine surgeons at 14 sites and randomized to spinal instrumentation with a low- or high-density screw pattern. Patients will return at 3-months, 1-year, and 2-years for exam, radiographs, and collection of patient-reported outcome scores. The Harms Study Group Foundation will serve as a collaborating organization and will provide database development and management, secure online data collection, centralized radiographic measurements, and data quality control. The University of Minnesota team will lead study design, protocol development, IRB/data use agreement contracts, patient randomization, and statistical analysis, including quarterly data review. Imaging will be obtained either with an EOS system or using a calibration belt during the radiographs, which allows for subsequent with the 3D modeling of the deformity. Six enrolling sites currently have this capability (EOS - Montreal, St. Louis, Iowa, Mayo, DuPont, and San Diego). An additional five sites already have calibration belts - Dallas, New York, Baltimore, Boston, U. of Rochester), and new calibration belts will be fabricated for the additional sites. The Montreal site will supervise collection of radiographic data with 3D capability and assist with troubleshooting and radiographic quality control. Although the study is primarily powered to detect change in percent correction of the major coronal curve, preliminary data will be gathered on axial and sagittal plane correction as well as complications, surgical factors, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥10 and ≤ 18 years
* Male or Female
* Diagnosis of idiopathic scoliosis for which surgery is recommended to prevent the curvature or to correct trunk disfigurement Lenke 1A curve pattern
* Curve cobb of 45° to 65°
* T5-T12 kyphosis measuring 0° to 40°
* Spina bifida Oculta is permitted
* Spondylolisthesis and Spondylolysis are permitted, as long as non- operative

Exclusion Criteria:

* Prior spinal surgery
* MRI abnormalities (including >4mm of Syrinx and/or Chiari malformation)
* Neuromuscular or other serious co-morbidities
* Thoracogenic or cardiogenic scoliosis
* Associated syndrome or developmental delay
* Unable or unwilling to firmly commit to returning for required follow-up

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-04-18 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Cobb Angle | pre-surgery ranging 1 year to 1 month and peri surgery at about 3-months, 1-year, and 2-year postoperative
  Radiographic, surgical, and patient-reported data will be gathered and analyzed to observe changes between time points. All radiographs will be taken with 3D analysis capability, either with a calibration belt using standard radiograph techniques or with an EOS imaging system. This will allow for additional detailed correction measures, such as change in spinal rotation (orientation of the planes of maximum curvature) and detailed coronal, sagittal and transverse plane measures. Bending films will be taken according to institutional protocol. The SRS-30, SAQ, and EQ5D will be collected at all clinical visits. Study questions will be aligned as much as possible with other prospective scoliosis protocols so as to minimize patient and surgeon response burden. The study protocol requires no additional visits or radiographs beyond standard of care.

SECONDARY OUTCOMES:
Blood Loss | During surgery, 1 time occurence
  Blood loss amount that occured during the surgical procedure.
Operative Time | 1 time measurement, occurs at surgery
  Length of time required to complete surgical procedure in either arm of the study (highest number or lowest number of screws).
3D parameter correction | collected during surgical procedure
  Surgeon reported measure of screw manipulation during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: David W Polly, MD, Principal Investigator — University of Minnesota
Locations (14):
- United States (13):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/ Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's Research Institute, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Washington University in St. Louis, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No